CLINICAL TRIAL: NCT05887934
Title: Investigation of Bone-Lead Level Associations With Brain and Mental Health and Treatment Response Among MUSC Psychiatry Patients
Brief Title: Bone-Lead Level Associations With Brain and Mental Health
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00126756
Record Dates: First submitted 2023-04-06; First posted 2023-06-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Lead Exposure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: X-Ray Fluorescence Analyzer — The XRF analyzer (the ThermoFisher Niton XL3t GOLDD+) is a portable x-ray fluorescent analyzer specifically configured to measure low levels of metals, lead in particular, in bone. The device is designed to rapidly assess cumulative lead exposure, not to support or sustain human life.

SUMMARY:
The goal of this study is to assess cumulative lead exposure among treatment-seeking patients in the MUSC hospital system receiving experimental transcranial magnetic stimulation (TMS), transcranial direct-current stimulation (tDCS), an electroencephalogram (EEG), and/or transcutaneous auricular vagus nerve stimulation (taVNS) therapies to determine whether lead exposure represents a risk factor for more severe mental illness or a modifier of treatment response. Information will be obtained from patients with a variety of neuropsychiatric disorders recruited to existing hospital studies. This information will include the results of bone-lead testing, brief cognitive tests, and self-reported psychiatric symptoms and behaviors.

DETAILED DESCRIPTION:
The goal of this study is to assess cumulative lead exposure among treatment-seeking patients in the MUSC hospital system receiving experimental transcranial magnetic stimulation (TMS), transcranial direct-current stimulation (tDCS), an electroencephalogram (EEG), and/or transcutaneous auricular vagus nerve stimulation (taVNS) therapies to determine whether lead exposure represents a risk factor for more severe mental illness or a modifier of treatment response. Information will be obtained from patients with a variety of neuropsychiatric disorders recruited to existing hospital studies. This information will include the results of bone-lead testing, brief cognitive tests, and self-reported psychiatric symptoms and behaviors. It is anticipated that the data will serve as preliminary data for research grant applications to support further data collection among a wider clinical and non-clinical population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Ability to read, write, and comprehend English
* Capacity to consent
* Consented for recontact, when applicable
* Negative pregnancy test

Additional inclusion criteria match those of parent studies, including:

* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in MPFC Theta Burst Stimulation as a Treatment Tool for Alcohol Use Disorder: Effects on Drinking and Incentive Salience (PRO 102709)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in An Open Label Study to Assess the Feasibility and Tolerability of Accelerated Theta Burst Repetitive Transcranial Magnetic Stimulation (iTBS-TMS) for the Treatment of Post-Partum Depression (PRO 73886)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in Developing a Novel rTMS Intervention for Transdiagnostic Psychosocial Rehabilitation: A Dose-finding Study (PRO 82315)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in Accelerated Repetitive TMS for Affective Dysfunction: Establishing the Dose-Response Curve (PRO 84111)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in Modeling and Modulating Mechanisms of Escape, Avoidance, and Approach in the Anxiety Disorder Spectrum (PRO 106843)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in Sign vs. Goal Tracking in Alcohol Use Disorder: Predicting problem alcohol use using a neurophysiological endophenotype of reward-based incentive salience attribution (PRO 124775)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in Transcranial Magnetic Stimulation and Decision Making (PRO 126644)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in The Influence of Mental States on Anticipation and Processing of Emotional Information (PRO 94001)
* Currently meets all inclusion criteria, has agreed to be recontacted, and has consented to participate in Optimizing Transdiagnostic Non-invasive Vagus Nerve Stimulation to Enhance Learning (PRO 107689)

Exclusion Criteria:

* Pregnant
* Current schizophrenia or psychotic disorder
* Inability or unwillingness of subject to give informed consent

Additional exclusion criteria match those of parent studies, including:

* Currently does not meet any exclusion criteria from MPFC Theta Burst Stimulation as a Treatment Tool for Alcohol Use Disorder: Effects on Drinking and Incentive Salience (PRO 102709)
* Currently does not meet any exclusion criteria from An Open Label Study to Assess the Feasibility and Tolerability of Accelerated Theta Burst Repetitive Transcranial Magnetic Stimulation (iTBS-TMS) for the Treatment of Post-Partum Depression (PRO 73886)
* Currently does not meet any exclusion criteria from Developing a Novel rTMS Intervention for Transdiagnostic Psychosocial Rehabilitation: A Dose-finding Study (PRO 82315)
* Currently does not meet any exclusion criteria from Accelerated Repetitive TMS for Affective Dysfunction: Establishing the Dose-Response Curve (PRO 84111)
* Currently does not meet any exclusion criteria from Modeling and Modulating Mechanisms of Escape, Avoidance, and Approach in the Anxiety Disorder Spectrum (PRO 106843)
* Currently does not meet any exclusion criteria from Sign vs. Goal Tracking in Alcohol Use Disorder: Predicting problem alcohol use using a neurophysiological endophenotype of reward-based incentive salience attribution (PRO 124775)
* Currently does not meet any exclusion criteria from Transcranial Magnetic Stimulation and Decision Making (PRO 126644)
* Currently does not meet any exclusion criteria from The Influence of Mental States on Anticipation and Processing of Emotional Information (PRO 94001)
* Currently does not meet any exclusion criteria from Optimizing Transdiagnostic Non-invasive Vagus Nerve Stimulation to Enhance Learning (PRO 107689)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The current study will recruit solely from research studies listed within the inclusion/exclusion criteria. The populations within the inclusion/exclusion criteria cover a wide range of psychiatric disorders including but not limited to alcohol use disorder (AUD), major depressive disorder (MDD), and anxiety spectrum disorders (ASD). There will be no exclusion based on gender or minority status. The investigators anticipate that at least 50% of the participants will be women. The percentage of minority participants is expected to be at least 5%. The investigators will make vigorous attempts to increase this number by posting advertisement flyers in minority communities.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Diagnoses | Baseline
  Count of participants varying neuropsychiatric disorders assessed by the Diagnostic Interview for Anxiety, Mood, and OCD and related Neuropsychiatric Disorders (DIAMOND)
Cognitive Function | Baseline
  Measurement of cognitive function as assessed by the Trail Making Test (TMT) as a way to assess central executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Kilpatrick, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No